CLINICAL TRIAL: NCT01343979
Title: Influenza A H1N1: Retrospective Analysis of PCR Confirmed Cases of H1N1 Infections in Styria - Risk Factors, Clinical Features and Outcome. Development of a Clinical Score for Suspected H1N1 Infection.
Brief Title: Influenza A H1N1: Retrospective Analysis of PCR Confirmed Cases of H1N1 Infections in Styria - Risk Factors, Clinical Features and Outcome.
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Robert Krause, MD, ao.Univ.Prof.Dr, Medical University of Graz
Other Study IDs: 23-049
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Clinically Suspected H1N1 Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- positive: Patients with clinically suspected H1N1 infection confirmed by positive H1N1 PCR
- negative: Patients with clinically suspected H1N1 infection and negative H1N1 PCR

SUMMARY:
This retrospective study will analyse all PCR-proven H1N1 cases from the influenza season 2009/2010 treated within the styrian "LKH hospital network". For this purpose all PCR-positive case files are reviewed in Medocs (electronic patients database) and data regarding clinical presentation, laboratory and radiological findings, treatment, outcome and preexisting underlying chronic illnesses will be systematically collected. In a second step the same data collection will be performed in a group of PCR-negative patients, which were tested during the influenza season 2009/2010 for influenza-like illness. The data from the PCR-positive group will be compared to the data from the PCR-negative group. We expect significant differences between the proven and unproven group regarding the primary presentation at hospital. Based on these results a clinical score will be developed. This score should improve H1N1 case identification in emergency departments, even if specific diagnostic test are negative (rapid antigen testing) or still pending (PCR), reduce the number of missed hospitalized H1N1 infection and optimize the decision making process in emergency departments regarding which patient has to be admitted with infection control measures and which not, and as infection control measures are expensive (face masks, gloves) and limited (isolation room), such a score should also reduce unnecessary expense. To evaluate the sensitivity and specificity of the score a prospective study will follow in the influenza season 2010/2011.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. All patients tested for influenza illness by PCR of respiratory tract specimens at the Institute of Hygiene, Karl-Franzens-University Graz, and at the Institute for Hospital Hygiene and Microbiology, KAGES Graz.
  2. Stratification according to the following definition:
* PCR-negative influenza-like illness (ILI) is defined as febrile illness tested by PCR for the presence of influenza infection but finally not proved as influenza infection.
* Influenza illness is defined as febrile illness confirmed by positive PCR as true influenza infection.

Exclusion Criteria:

* NONE

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients tested for influenza illness by PCR of respiratory tract specimens at the Institute of Hygiene, Karl-Franzens-University Graz, and at the Institute for Hospital Hygiene and Microbiology, KAGES Graz.
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
clinical presentation of H1N1 compared to other viral infections | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hoenigl, MD, Principal Investigator — Medical University of Graz; Robert Krause, MD, Principal Investigator — Medical University of Graz; Holger Flick, MD, Principal Investigator — Medical University Hospital Graz
Locations (1):
- Medical University Hospital of Graz, Graz, Styria, Austria